CLINICAL TRIAL: NCT00077519
Title: A Phase I Trial of the Farnesyltransferase Inhibitor, R115777 (NSC# 702818) and Radiotherapy in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Tipifarnib and Radiation Therapy in Treating Patients With Unresectable Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: UPCC 20203; CDR0000352182; NCI-6407
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tipifarnib; Radiotherapy

INTERVENTIONS:
Drug: tipifarnib
Radiation: radiation therapy

SUMMARY:
RATIONALE: Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for their growth and may make them more sensitive to radiation therapy. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving tipifarnib together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of tipifarnib when given together with radiation therapy in treating patients with unresectable locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and dose-limiting toxic effects of tipifarnib when administered with radiotherapy in patients with unresectable locally advanced pancreatic cancer.

Secondary

* Determine the 3-month clinical response in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of tipifarnib.

Patients receive oral tipifarnib once or twice daily on weeks 1-8. Patients also undergo concurrent radiotherapy daily, 5 days a week, on weeks 2-8.

Cohorts of 3-6 patients receive escalating doses of tipifarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 1, 3, and 6 months.

PROJECTED ACCRUAL: A total of 8-18 patients will be accrued for this study within 12-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed pancreatic cancer

  * Locally advanced disease
* Unresectable disease requiring radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* AST or ALT < grade 2 elevation
* Bilirubin ≤ 2.0 mg/dL* NOTE: *Prior biliary stent procedure to normalize bilirubin levels allowed

Renal

* Creatinine ≤ 1.5 times normal

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No peripheral neuropathy ≥ grade 2
* No known allergy to imidazole drugs, including any of the following:

  * Clotrimazole
  * Ketoconazole
  * Miconazole
  * Econazole
  * Fenticonazole
  * Isoconazole
  * Sulconazole
  * Tioconazole
  * Terconazole

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior experimental or standard chemotherapy and recovered
* No concurrent experimental chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior upper abdominal radiotherapy

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2004-01; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Michael Hahn, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States